CLINICAL TRIAL: NCT01504945
Title: Red Blood Cell Transfusion in Patients With Acute and Chronic Coronary Syndrome
Brief Title: Red Blood Cell Transfusion in Patients With Coronary Artery Disease (CAD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2009P000436
Record Dates: First submitted 2011-04-25; First posted 2012-01-06 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Acute Coronary Syndrome; Anemia
Keywords: chronic coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Anemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RBC transfusion (Active Comparator)
  Interventions: Other: RBC transfusion
- Normal saline infusion (Placebo Comparator)
  Interventions: Other: Normal saline infusion

INTERVENTIONS:
Other: RBC transfusion — 1 bag of packed red blood cells
  Arms: RBC transfusion
Other: Normal saline infusion — 500 mL of normal saline infusion
  Arms: Normal saline infusion

SUMMARY:
Patients with a low blood count (anemia) with stable or unstable coronary artery disease consistently show worse clinical outcomes. It is unclear whether this association is confounded since anemic patients tend to be also sicker i.e. have lower ejection fractions or more comorbidities and this would be the reason for the worse outcomes rather than anemia. The coronary arteries are a unique vascular bed insofar that across the cardiac circulation oxygen extraction is close to maximal at rest. Thus increases in demand can only be met by increases in blood flow and hemoglobin concentration since oxygen extraction is maximal at rest. It is natural to assume that maximization of oxygen delivery in the setting of active coronary syndrome (ACS) is beneficial to the patient since oxygen extraction and coronary blood flow is fixed. In fact, in most intensive care units patients with ACS are transfused to a HCT of 30%. However, retrospective analysis of trial data showed at best mixed results in clinical outcome when patients with ACS were transfused and in fact in some studies showed consistently worse outcomes than non-transfused patients. Similar disappointing results have recently published in patient who underwent coronary artery bypass grafting (CABG).

This study is designed to determine the effect of red blood cell (RBC) transfusion on oxygen consumption, cardiac, microcirculatory and endothelial function in patients with active coronary artery disease. For this study active coronary artery disease will be defined as the patient having undergone within the past 4 days of recruitment either a myocardial infarction due to atherothrombosis (AHA type I myocardial infarction) or surgery for coronary artery bypass grafting.

In specific this study will test the hypothesis whether RBC transfusions improves cardiac and vascular function in patients with a hematocrit of less than 30% with active coronary artery disease.

Aims of this study are to determine whether RBC transfusion in patients with active coronary artery disease and anemia:

* increases oxygen delivery to the peripheral tissues.
* increases whole-body oxygen consumption.
* decreases nitric oxide bioavailability, endothelial, microcirculatory, and myocardial function, and/or increases platelet aggregation

DETAILED DESCRIPTION:
Adverse clinical outcomes are reduced when critically ill patients are only transfused if their hematocrit drops below 21%: Hematocrit (HCT) is a measure of the severity of anemia. A HCT is considered normal if it ranges between 38 and 48% of total blood volume. In critically ill patients anemia is very common; about 95% of patients admitted to the intensive care unit have hemoglobin levels below normal by intensive care unit (ICU) day 3.{Corwin, 1995 #8809;Rodriguez, 2001 #8810} The transfusion trigger of "30/10" (HCT < 30%, hemoglobin <10 g/dl) has been suggested in a case series of trauma patients as early as 1942.{Adam, 1942 #8811} Since then these triggers have largely been a matter of faith, without prospective data supporting an improvement in clinical outcome. Several clinical trials conducted in the past two decades have shown at least equivalence in clinical outcomes when a more conservative transfusion trigger of hemoglobin 7-9 g/dL is applied to a critically-ill patient population.{Hebert, 1999 #8812;Vincent, 2002 #8814;Corwin, 2004 #8813} The transfusion trigger in patients with acute coronary syndrome (ACS) or recent coronary artery bypass grafting as a subset of critically ill patients is more controversial, and in most intensive care units a more liberal approach to transfusions for these patients is typically chosen.{Gerber, 2008 #8815} However, the efficacy of RBC transfusion appears to be significantly more limited than empirically assumed in patients with active coronary artery disease. The TRICC investigators performed a subset analysis and independent study of their patient cohort of critically-ill patients with cardiovascular disease.{Hebert, 1997 #8835} They found that a transfusion hemoglobin trigger of 7 g/dL is safe. Furthermore, greater end-organ dysfunction was recorded in patients with a liberal transfusion trigger, and the overall mortality was similar between the study cohorts for any time interval (intensive care unit, over the course of hospital stay, at 30-d and 60-d follow-up).{Hebert, 1999 #8812}

ACS patients should receive a transfusion if their HCT is less than 24%: Several retrospective studies have shown that in general, transfusion of RBC in patients with ACS and a hematocrit > 24% is neutral or very slightly beneficial and causes harm if HCT > 30%. {Rao, 2004 #8836;Yang, 2005 #8837;Sabatine, 2005 #8827;Singla, 2007 #8838;Singla, 2007 #8838} Such small (if any) benefit is not intuitive, in light of an increase in arterial oxygen content by a PRBC transfusion and therefore decrease in cardiac output and oxygen consumption. Two very beneficial effects in patients with active coronary artery disease. Indeed, increasing arterial oxygen content by transfusion may either 1) not increase oxygen delivery to the myocardium distal to an anatomic coronary stenosis or 2) have other deleterious biological effects on the cardiovascular system. Despite the results that RBC transfusion in unstable coronary artery disease has very little beneficial effects, most clinicians (standard of care) transfuse patients with ACS to a HCT of 30% regardless of potential adverse side effects of RBC transfusions. The guidelines for transfusion practice at the BIDMC for instance differentiate between hemodynamically stable and bleeding patients. The HCT of bleeding patients should be greater then 30%. In hemodynamically stable patient they further differentiate between patients with and without signs of end-organ ischemia. In patients without end-organ ischemia a HCT of 21% is tolerated and in patients with end-organ ischemia such as active coronary artery disease the HCT should be > 30%.

Storage of RBC before transfusion lowers the function of the RBCs: In a retrospective study in patients undergoing coronary artery bypass grafting (CABG) a recent study found that RBC transfusions were associated with an increased risk of mortality and short term and long term postoperative complications when patients were transfused with stored RBCs (older than 14 days). This association remained significant even after controlling for the assumption that patients receiving blood transfusions are in general sicker and therefore more prone to complications.{Koch, 2008 #8847} Since the introduction of acid-citrate-dextrose as a preservative it was possible to store blood for several weeks currently up to 42 days. The criteria for the decision when is blood storage too long is based arbitrarily on red blood cell survival in the recipient after 24 hours and should be greater than 70%.{Mollison, 1942 #8848} In the past decades however it has been established that transfused and surviving red blood cells exhibit quite different physiologic properties when compared to native RBCs. This phenomenon is called the storage lesion. There is a rapid depletion of 2,3 diglycerophosphate (2,3-DPG) with storage.{Bunn, 1968 #8849} This has a profound impact on hemoglobin affinity reducing oxygen release from hemoglobin by as much as 25% at similar change in oxygen saturation. Of note within 72h about 50% of the 2,3-DPG is restored in the transfused RBCs. Moreover, there is a marked decrease of adenosine triphosphate (ATP), which reduces deformability of transfused RBCs and the ability of the RBCs to navigate the microcirculation.{Dern, 1967 #8850}

Infusion of stored RBCs causes hemolysis which in turn reduces nitric oxide bioavailability: Significant hemolysis (a condition in which RBC burst and the contents of RBC leak outside; in particular free hemoglobin) occurs both during storage and in particular during transfusion.{Sowemimo-Coker, 2002 #8851} Free hemoglobin outside of RBCs scavenges nitric oxide. Nitric oxide (NO) is a colorless gas, which is produced by the inner lining of the vessels (endothelium). It acts as D5W lubricant for vessels. It keeps blood vessels open and "lubricates them" so blood cell can flow through these blood vessels more easily. A decrease in nitric oxide bioavailability causes vasoconstriction and increased RBC adhesion to endothelium which in turn decreases microcirculatory flow.{Reiter, 2002 #6096} RBCs also contain arginase which released into the circulation will further enhance nitric oxide depletion by reducing its precursor arginine.{Kato, 2005 #7955}

The investigators will systematically examine the effects of RBC transfusion on systemic oxygen delivery, whole body oxygen consumption, nitric oxide bioavailability, endothelial function, cardiac performance, microcirculatory function, and platelet aggregation in patients with active coronary artery disease, presenting to the BIDMC with anemia, defined as hematocrit of < 30%. This is to test our hypothesis that depletion of the nitric oxide pool by transfusion-associated hemolysis causes a decrease in microcirculation, endothelial, and platelet function. To the best of our knowledge there is no study to date that explores the physiologic effects of RBC transfusion in patients with active coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* ACS as defined by a patient who has cardiac chest discomfort and a troponin (cTnT) elevation of greater than 0.1 ng/mL.
* Pt. who is s/p CABG
* Patients with chronic coronary artery disease will be recruited as defined as past history of myocardial infarction, percutaneous coronary intervention, CABG, or history of coronary artery disease documented in the medical record.
* Anemia as defined by HCT between 21%-30%.

Exclusion Criteria:

* Patients with stage III/IV heart failure
* Patients who are actively bleeding requiring immediate transfusion.
* Pregnant patients will be excluded.
* Patients taking sildenafil (Viagra) or other drugs like it, such as vardenafil (Levitra), or tadalafil (Cialis) within 48 hours before the study.
* Patients on iv nitroglycerine infusion.
* Patients who present with ACS or CABG surgery and who are hemodynamically unstable or require immediate revascularization.
* Patients who have received a blood transfusion 24 hours prior to the start of the study.
* Patients with a HCT of < 21% and those that have chest tube drainage greater then 30 mL/h will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function as measured by flow mediated dilation | within 1 day of transfusion

SECONDARY OUTCOMES:
platelet function | within one hour of transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Andre Dejam, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States